CLINICAL TRIAL: NCT02359721
Title: Efficacy of Clarithromycin is an Adjunct to Scaling and Root Planing .A Clinical Microbiological and Immunological Study.
Brief Title: Clarithromycin is an Adjunct to Scaling and Root Planing
Acronym: CASRCMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, J.surya prasanna, DR.J. SURYA PRASANNA, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RADHIKA DISSERTATION
Record Dates: First submitted 2015-01-05; First posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-01

CONDITIONS: Periodontitis
Keywords: Colony forming units Antimicrobial agents; Microbial colonization
MeSH Terms: conditions — Periodontitis; Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- test group (Experimental): Base line scaling and root planing was done. Clarithromycin tablet 500 mg( Clarino-500) was given for a period of 7 days orally two times per day
  Interventions: Drug: tablet clarithromycin 500 mg (Clarino-500) orally
- control (No Intervention): scaling and root planing

INTERVENTIONS:
Drug: tablet clarithromycin 500 mg (Clarino-500) orally — orally
  Other Names: Clarino-500
  Arms: test group

SUMMARY:
The present study was done to evaluate the effect of clarithromycin as an adjunct to scaling and root planning at baseline, three months and six months intervals . Clinical, microbiological and immunological parameters were taken. Clinical parameters include gingival index , probing depth and clinical attachment level. In the present study, improved clinical and microbiological outcomes were attained using adjunctive clarithromycin, including GI, PD reduction, CAL gain and reductions in the frequency of detection of C-reactive protein, Pg, Aa. These results together with the recommended easy dosage and limited side effects make the use of this antibiotic in the treatment of periodontitis patients but only for a shorter period of time.

DETAILED DESCRIPTION:
Background & Objectives: Along with conventional non-surgical periodontal therapy (NSPT) systemic antimicrobials may provide more effective treatment for chronic periodontitis by targeting tissue-invasive bacteria. The aim of this study was to evaluate the adjunctive effects of oral clarithromycin (CLM) to nonsurgical periodontal therapy for chronic periodontitis.

Materials and Methods: 30 patients were categorized into two groups: test group - Base line scaling and root planing(SRP) was done. Clarithromycin tablet 500 mg( Clarino-500) was given for a period of 7 days orally two times per day. control group -only SRP done . Clinical parameters were recorded at baseline , 3 months, and six months interval .They included gingival index (GI), probing depth (PD), and clinical attachment level (CAL). Also microbial analysis of subgingival plaque samples was done at baseline, 3months and six months interval to estimate the levels of Pg and Aa bacteria using culture methods. Immunological parameter like estimation of C-Reactive protein was done in both groups at baseline 3 months and 6 months period. tests were used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ranged between 30- 50 years with chronic periodontitis
* Patients with Probing Depth (PD)- >5mm, Clinical Attachment Level( CAL)- >3mm
* Systemically healthy individuals

Exclusion Criteria:

* Patients below the age of 30 years
* Patients who have undergone periodontal therapy 3 months prior to study
* Active /passive smokers
* Any antibiotic use 3 months prior to study
* Pregnant women and lactating mothers
* Un co- operative/ retarded patients
* Drug allergy/ other allergies
* Any systemic diseases

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of Clarithromycin, as measured by reduction Gingival bleeding | 6 months
  0,3,6 months
Efficacy of Clarithromycin, as measured by Pocket probing depth | 6 months
Efficacy of Clarithromycin, as measured by Clinical attachment gain | 6 months
c-reactive protein levels | 6 months
Pg and Aa bacterial count | 6 months

REFERENCES:
- [Background] Kathariya R, Pradeep AR, Raghavendra NM, Gaikwad R. Evaluation of subgingivally delivered 0.5% clarithromycin as an adjunct to nonsurgical mechanotherapy in the management of chronic periodontitis: a short-term double blinded randomized control trial. J Investig Clin Dent. 2014 Feb;5(1):23-31. doi: 10.1111/jicd.12009. Epub 2012 Oct 25. PMID 23097216
- [Background] Bajaj P, Pradeep AR, Agarwal E, Kumari M, Naik SB. Locally delivered 0.5% clarithromycin, as an adjunct to nonsurgical treatment in chronic periodontitis with well-controlled type 2 diabetes: a randomized controlled clinical trial. J Investig Clin Dent. 2012 Nov;3(4):276-83. doi: 10.1111/j.2041-1626.2012.00168.x. Epub 2012 Sep 13. PMID 22976782
- [Background] Agarwal E, Pradeep AR, Bajaj P, Naik SB. Efficacy of local drug delivery of 0.5% clarithromycin gel as an adjunct to non-surgical periodontal therapy in the treatment of current smokers with chronic periodontitis: a randomized controlled clinical trial. J Periodontol. 2012 Sep;83(9):1155-63. doi: 10.1902/jop.2012.110600. Epub 2012 Jan 16. PMID 22248223
- [Result] Raghunatha K, George JP. Periodontal tissue and serum concentration of clarithromycin after systemic administration in patients affected by chronic periodontitis. J Periodontol. 2013 Sep;84(9):e17-22. doi: 10.1902/jop.2013.120521. Epub 2013 Mar 1. PMID 23451987
- [Result] Pradeep AR, Kathariya R. Clarithromycin, as an adjunct to non surgical periodontal therapy for chronic periodontitis: a double blinded, placebo controlled, randomized clinical trial. Arch Oral Biol. 2011 Oct;56(10):1112-9. doi: 10.1016/j.archoralbio.2011.03.021. Epub 2011 May 6. PMID 21529775
- [Result] Burrell RC, Walters JD. Distribution of systemic clarithromycin to gingiva. J Periodontol. 2008 Sep;79(9):1712-8. doi: 10.1902/jop.2008.080013. PMID 18771373
- [Result] Piccolomini R, Catamo G, Di Bonaventura G. Bacteriostatic and bactericidal in vitro activities of clarithromycin and erythromycin against periodontopathic Actinobacillus actinomycetemcomitans. Antimicrob Agents Chemother. 1998 Nov;42(11):3000-1. doi: 10.1128/AAC.42.11.3000. PMID 9797240